CLINICAL TRIAL: NCT00482859
Title: Sleep Disturbance and Sleep Quality in Women With Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Suzette L. Sewell Scheuermann RN, University of Kentucky College of Nursing
Other Study IDs: 07-0188-P2G; Non-Applicable
Record Dates: First submitted 2007-06-03; First posted 2007-06-05 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this week long study is to describe sleep and problems with sleep in women diagnosed with Fibromyalgia syndrome.

DETAILED DESCRIPTION:
At least 50 women over 18 years of age are invited to volunteer in this study. Sleep quality and problems with sleep will be described using several kinds of measures. Questionnaires on sleep and Fibromyalgia will be completed by the volunteer. In addition, the volunteer will complete a sleep diary for at least 7 days and wear an Actiwatch (a wrist watch like device that measures sleep). At completion of the study, participants will be provided a print out of their sleep obtained from the Actiwatch.

Participants may not be in the study if they work night shift (11 pm - 7 am) or have been diagnosed with a condition called sleep apnea.

Participants need not live in Kentucky to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old; diagnosed with Fibromyalgia;

Exclusion Criteria:

* Volunteer works night shift (11PM - 7AM);
* Volunteer has been diagnosed with sleep apnea.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with Fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzette L Sewell, RN MSN, Principal Investigator — University of Kentucky